CLINICAL TRIAL: NCT03396848
Title: An Online Sexual Health and Rehabilitation eClinic (SHAReClinic) for Prostate Cancer Patients and Their Partners: a Feasibility Study
Brief Title: Sexual Health and Rehabilitation eClinic (SHAReClinic)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Tom Baker Cancer Centre (Other); Vancouver Coastal Health (Other Government); Sunnybrook Health Sciences Centre (Other); Nova Scotia Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHAReClinic 001
Record Dates: First submitted 2017-12-12; First posted 2018-01-11 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer; Sexual Dysfunction
Keywords: Rehabilitation; Online Clinic
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Patient will have access to an online clinic after their prostate cancer treatment. This is a feasibility study to determine whether it would be feasible to implement SHAReClinic as a pan-Canadian sexual health and rehabilitation intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHAReClinic (Experimental): All participants will have access to the online clinic
  Interventions: Other: SHAReClinic

INTERVENTIONS:
Other: SHAReClinic — Online clinic with educational modules

SUMMARY:
In addressing the need for effective post treatment support for men (and their partners) following treatment for prostate cancer, the investigators will employ an innovative SHAReClinic (Sexual health and Rehabilitation eClinic Program) that emphasizes: 1) a bio-medical component (erectile rehabilitation), focused on the long term return of erectile functioning firm enough for penetration with or without erectile agents/devices; and 2) a psychological component (intimacy maintenance), involving the maintenance or restoration of couples' intimacy. Through comparison research, the eClinic will be analyzed and made comparable in quality to the programs offered currently at leading institutions in major metropolitan areas, thus providing personalized, comprehensive cancer care to all Canadians.

DETAILED DESCRIPTION:
The considerable prevalence of sexual dysfunction (SD) after prostate cancer treatment, coupled with the severity/breadth of impact and lack of successful intervention makes SD post-treatment one of the most substantial health-related quality of life burdens in all of cancer survivorship. In 2014, it is estimated that 24,000 Canadians will be diagnosed with prostate cancer (PC) and 4,100 men will die of the disease. Accordingly, 19,900 men will be added to the pool of Canadian prostate cancer survivors in just one year. Today, there are approximately 250,000 prostate cancer survivors across Canada. Research with men in post-radiation therapy indicates that 24-59% suffer SD, while 40%-75% of men in post-radical prostatectomy suffer SD. Sixty percent of men experience significant distress in response to SD. Distress is especially elevated in younger men and evidence suggests that partners may experience even greater distress than patients. Research examining the nature of the distress reveals that the significance of SD reaches far beyond the ability to have an erection, and resides in its complex psychosocial implications, including intimacy loss, low self-esteem, guilt, depression, anxiety, and anger. Additional evidence suggests that patients' SD-related distress can lead to long-term maladjustment in their overall relationships with their partners. The burden of SD following treatment for prostate cancer is responsible for the single greatest impact on patient/partner/couple health-related quality of life; substantially more so than concern for cancer recurrence. Unfortunately, there are no reported interventions to date that have been successful in reducing the impact of SD following treatment, on long-term couple health-related quality of life. Accordingly, given the extensive impact of SD on patient/partner health-related quality of life (HRQOL) there is an existent need for restorative/rehabilitative intervention.

The current study proposes the application of an online bio-psychosocial intervention to address sexual dysfunction following treatment for prostate cancer. The bio-medical approach will apply a broader definition of penile rehabilitation which will focus on applying a systematic pro-erectile aid regimen to assist patients in achieving long-term return of erectile functioning, firm enough for penetration, with or without the use of pro-erectile agents/devices. The investigators have termed this bio-medical rehabilitation approach, Erectile Rehabilitation. As such, the rehabilitation algorithm includes but is not limited to the goal of return of natural functioning. Overall, the investigators endeavour to help patients find and adapt to the least invasive pro-erectile agent /device that is successful in achieving desired erections. The investigators justify this approach through extensive research that demonstrates that, following prostate cancer treatment, patients who use pro-erectile agents report better erectile functioning versus those who do not use pro-erectile agents. In addition to addressing Erectile Rehabilitation, this intervention will offer psychosocial support, with the goal of helping couples maintain or restore intimacy after treatment for prostate cancer. Health coach interventions aim at improving sexual satisfaction following prostate cancer treatment have been shown to improve distress and sexual function, and provide patients with the information on pro-erectile aids and couples' experiences.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following inclusion criteria will be eligible for the study:

* Men who are scheduled for a RP (open, robotic) for the first-line treatment for localized prostate cancer;
* Men who are scheduled for Radiation treatment (brachytherapy, external beam) for localized prostate cancer as their first line of treatment
* Men who are hormone and/or chemotherapy-naïve
* Men who have access a computer with internet access
* Men who are 18 years of age or older

OR:

• Partners of men who meet the above criteria and are 18 years of age or older

Exclusion Criteria:

Patients/couples will be excluded from study participation if:

* the patient or partner lacks English proficiency
* the patient is on nitrate therapy or has other contra-indications to phosphodiesterase type 5 inhibitors (PDE5i's)
* the patient or partner has a medical condition that would preclude safe sexual activity
* the patient has had previous treatment for PC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of relationship and Intimacy from different time points | This questionnaire will be completed by coupled participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Miller Social Intimacy Scale (MSIS):MSIS is a 17-item measure of the maximum level of intimacy currently experienced is used in this study. Each question has a scale of 1-10 with a higher score representing higher level of intimacy.
Change of Relationship and Intimacy for male participants from different time points | This questionnaire will be completed by male participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  The Sexual Health Inventory for Men (SHIM): SHIM was developed and validated as a brief, easily administered, patient-reported diagnostic tool for men as a measure for male optimal sexual health for Bio-medical Responders and Bio-medical Non-Responders. SHIM has 5 items in all with a scale from 0(1) to 5. Higher number indicates a better sexual function.
Change of Relationship and Intimacy for female participants from different time points | This questionnaire will be completed by female participants at T1 (pre-treatment online visit), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment)
  Female Sexual Function Inventory (FSFI): the FSFI is a brief, 19-item self-report measure of female sexual function that provides scores on six domains of sexual function (Desire, Arousal, Lubrication, Orgasm, Satisfaction, Pain) as well as a total score. The full scale score is obtained by adding the six domain scores. It should be noted that within the individual domains, a domain score of zero indicates that no sexual activity was reported during the past month. Higher score indicates a better sexual function.
Change of sexual function from different time points | This questionnaire will be completed by all participants at T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Prolonged Grief about the Loss of Sexual Function (PGLSF) is adapted from Prigerson's measure of prolonged grief in bereavement. Combinatoric analyses identified the most sensitive and specific Prolonged Grief Disorder (PGD) algorithm that was then tested to evaluate its psychometric validity. Criteria require reactions to a significant loss that involve the experience of yearning (e.g., physical or emotional suffering as a result of the desired, but unfulfilled, reunion with the deceased) and at least five of the following nine symptoms experienced at least daily or to a disabling degree: feeling emotionally numb, stunned, or that life is meaningless; experiencing mistrust; bitterness over the loss; difficulty accepting the loss; identity confusion; avoidance of the reality of the loss; or difficulty moving on with life. The PGLSf consists of 22 items with a Likert scale of 1 to 5: higher score indicates a higher grief level.
Change of Sexual desire and activity from different time points | This questionnaire will be completed by all participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Sexual Interest and sexual activity are used were to measure sexual activity and sexual desire in this study. For patients with cancer who may or may not have sexual dysfunction, the PROMIS SexFS measures provide a comprehensive assessment of key domains of sexual function and satisfaction. The questionnaire has 13 items in total with Likert scale of 1 to 5. Higher score indicates a higher sexual activity/desire level.
Change of psychological stress from different time points | This questionnaire will be completed by all participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Hospital Anxiety and Depression Scale (HADS) is used to determine the levels of anxiety and depression that participants are experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each question has a scale of 0 to 3 and the total score can be calculated for the two domains (anxiety and depression) by adding the scores together. For each domain, a score of 0-7 = Normal level of anxiety/depression; a score of 8-10 = borderline case of anxiety/depression; 11-21 = case of anxiety/depression.
Change of Sexual Distress from different time points | This questionnaire will be completed by all participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Sexual Distress Scale (SDS) is used in this study to measure sexual distress. SDS was created and validated to assess sexually related distress-that is, distress associated with inadequate or impaired sexual function. It has 13 items in all with a Likert scale from 0 to 4; higher score indicates a higher distress level.
Change of prostate cancer- related Quality of Life from different time points | This questionnaire will be completed by patient-participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  Patient Oriented Prostate Cancer Utility Survey (PORPUS) was used in this study to measure quality of life for patients after prostate treatment. The PORPUS contains 10 questions. There are 5 general questions (pain, energy, emotional well-being, social well-being, and relationship with physician) and 5 prostate cancer-specific questions (sexual function and desire, urinary frequency and incontinence, and bowel function), each with four to six possible answers, scoring 1 to 4 (6). Higher score indicates a better function in the respective domain.
Change of prostate cancer- related Quality of Life from different time points (expanded) | This questionnaire will be completed by patient-participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online clinic visits.
  Expanded Prostate Cancer Index Composite (EPIC) is used in this study: EPIC is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. The version we used contains 26 item and the 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-itemscale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL (Health-Related Quality of Life).
Change of general Quality of Life from different time points | This questionnaire will be completed by all participants at T1 (pre-treatment), T2 (6 weeks after treatment), T5 (6 months after treatment) and T6 (12 months after treatment) online visits.
  EQ-5D Health Questionnaire is used in this study as a standardized instrument to measure of health-related quality of life. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each item has 3 levels of severity with a higher number indicating better quality of life.

SECONDARY OUTCOMES:
Demographic Information | This questionnaire will be completed by all participants at T1 (pre-treatment) online visit
  Demographic Questionnaire will be used to collect social-demographic information from participants for analysis.
Satisfaction to the program | This questionnaire will be completed by all participants at T6 online visit (12 months after treatment).
  Satisfaction Questionnaire was used to receive participants' feedback on the website and their experience with the online clinic visits. The questionnaire contains 29 items in 4 domains: Satisfaction with SHAReClinic Program Referral, Registration & Onboarding; Satisfaction with Online SHAReClinic Portal and Content (Educational Modules); Satisfaction with SHAReClinic Health Coach and Overall Satisfaction with SHAReClinic Program. A Likert Scale of 1 to 5 is used for the items with a higher score indicating better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Matthew, PhD, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
The study data will be shared via an academic publication